CLINICAL TRIAL: NCT03183635
Title: A Randomized Controlled Trial of Rapid Movement Therapy With Real-time Feedback to Improve Balance Recovery for Fall Prevention After Stroke
Brief Title: Rapid Movement Therapy for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12131911
Record Dates: First submitted 2016-09-14; First posted 2017-06-12 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect based Rapid Movement Therapy (Experimental): Kinect based Rapid Movement Therapy (RMT) training requires participants to move their limbs very rapidly to reach-to-grasp or step towards a virtual target appear suddenly on a screen, which is designed to their range of motion as well as response speed.
  Interventions: Procedure: Balance training
- Conventional balance training (Placebo Comparator): Conventional balance training involves some slow and low-impact muscle strengthening and mobilizing exercises.
  Interventions: Procedure: Balance training

INTERVENTIONS:
Procedure: Balance training — Improvement of balance ability in stroke patients

SUMMARY:
Stroke survivors have higher risks of falling compared to other healthy non-stroke adults. Stroke patients' balance can be trained by Kinect-based training that enable user friendly and interactive training.

ELIGIBILITY:
Inclusion Criteria:

1. have single stroke with onset >1 year,
2. have unilateral paresis,
3. are 50 years of age or older,
4. able to stand without aid for at least 15min,
5. have moderate level of motor impairment in the affective upper limb, i.e. 15≤ Fugl-Meyer Assessment for upper-extremity(FMA-UE) ≤ 45,
6. have some level of deficit in balance control, i.e. Berg Balance Scale(BBS)< 52/56,
7. have a minimum Snellen visual acuity of 20/40 with/without spectacles,
8. have a minimum Mini-Mental-Status-Examination score of 22/30, and
9. have to be able to follow the training procedures.

Exclusion Criteria:

1. enrolled in other rehabilitation program in the study duration,
2. have other neurological conditions in addition to stroke (e.g. Parkinson's disease),
3. have unstable cardiovascular disease (e.g. history of heart disease, or poorly controlled hypertension, i.e. blood pressure >160mmHg/100mmHg), or
4. have other serious diseases or conditions (e.g. osteoporosis, recent joint replacement surgery, amputation) that preclude them from participating in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 3-month follow-up
  A 14-item objective measure designed to assess static balance and fall risk in adult populations
Timed Up and Go (TUG) | 3-month follow-up
  It is used to assess mobility, balance, walking ability, and fall risk in older adults

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) of Motor Recovery after Stroke | 3-month follow-up
  It is used to evaluate and measure recovery in post-stroke hemiplegic patients
Activities-specific Balance Confidence (ABC) Scale | 3-month follow-up
  Subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness
Barthel Index of Activities of Daily Living | 3-month follow-up
  It is used to assess the ability of an individual with a neuromuscular or musculoskeletal disorder to care for him/herself
Electromyography (EMG) | 3-month follow-up
  It is used to detect the muscle activity
"lean-and-release" postural system | 3-month follow-up
  It is used to evaluate balance-recovery in chronic stroke patients. Participants will wear a safety harness designed to prevent impact between body and floor, and they will be asked to stand on two force plates in standardized stance and lean forward with around 10% body weight supported by a cable attached to a release mechanism. Compensatory balance-recovery reactions will be evoked by the sudden release of the support cable, inducing a forward fall. Participants will be evaluated under three different conditions: no handrail, handrail on the unaffected side, and handrail on the affected side.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Junata M, Cheng KC, Man HS, Lai CW, Soo YO, Tong RK. Kinect-based rapid movement training to improve balance recovery for stroke fall prevention: a randomized controlled trial. J Neuroeng Rehabil. 2021 Oct 11;18(1):150. doi: 10.1186/s12984-021-00922-3. PMID 34635141